CLINICAL TRIAL: NCT04263311
Title: Scaling Community-Clinical Linkage Models to Address Diabetes and Hypertension Disparities in the Southeast United States
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-01192
Record Dates: First submitted 2020-01-31; First posted 2020-02-10 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Health Workers (CHW) treatment group (Experimental): Once recruited and consented, surveys will be administered and collected at baseline and 6 months in person or by a study coordinator within two weeks of completion of the CHW coaching component of the intervention. Participants enrolled in the intervention will receive monthly text and phone call reminders. in addition, multiple sessions will be hosted at varying times/days of the week to accommodate schedules of both working individuals and at-home caretakers. Finally, small incentives will be provided at each session to encourage ongoing attendance, and a cash raffle prize will be distributed at program completion for individuals who attend all five sessions.
  Interventions: Behavioral: CHW
- Control group (No Intervention): Control participants will be offered the health education sessions as a point of service and not for research purposes

INTERVENTIONS:
Behavioral: CHW — Participants will undergo 5 group-based health education sessions on hypertension and diabetes management and provide culturally and linguistically tailored health information and resources There will be 2 one-on-one in-person meetings and up to 7 follow-up calls/meetings to engage in goal-setting activities regarding changes to health behaviors, medication adherence, or other issues related to diabetes prevention as identified jointly by patient and CHW. Participants will develop with the CHW and receive a copy of their long-term and short-term Participant Action Plan. Referrals to other services available in the community (i.e. exercise classes, social services, mental health, tobacco cessation, etc.
  Arms: Community Health Workers (CHW) treatment group

SUMMARY:
The purpose of this study is to work with primary care physicians and their staff, and with community health workers (CHWs) to improve diabetes and hypertension management, health behaviors and improve blood pressure for South Asian patients with uncontrolled diabetes and hypertension in primary care clinics in Atlanta, Georgia. The CHWs are community members who are trained to work with patients to address health needs holistically by providing information on wellness, nutrition, stress relief, and blood pressure management in a culturally-appropriate and language-appropriate manner.

DETAILED DESCRIPTION:
The study will provide research training, technical assistance, and capacity-building to community and clinical sites in Georgia for implementation of culturally tailored, evidenced-based CHW programs to improve HTN and diabetes management for South Asians. In addition, the use a multi-theoretical framework to test the effectiveness of a CHW-led intervention compared to usual care among South Asian individuals with diabetes and uncontrolled HTN in Atlanta. The primary outcome is blood pressure control, defined as 130/80 mmHg. It is hypothesized that, compared to usual care, individuals receiving the CHW intervention will be 20% more likely to achieve blood pressure control at 6 months.

And to apply RE-AIM and CFIR frameworks to delineate factors influencing appropriateness, fidelity, adoption, and maintenance of the intervention within clinical and community settings to optimize intervention replication.

In addition, this study will serve as a national information and dissemination resource in the adaptation of evidence-based strategies to reduce geographic disparities in HTN and diabetes across Asian American groups.

ELIGIBILITY:
CHW intervention:

Inclusion Criteria:

* identified as of South Asian ethnicity
* are at least 21 years of age and younger than age 80
* had an appointment with a physician or mid-level clinician for routine non-emergent primary care in the last 12 months
* a diagnosis of diabetes
* a diagnosis of hypertension
* an uncontrolled BP reading (>130/80mmHg) in the last 6 months

Provider Surveys Inclusion criteria

* clinicians employed by the clinic
* have enrolled into the study.

Key Informant Interviews Inclusion criteria

* must be a provider, clinic manager, or community health worker.

CHW intervention

Exclusion Criteria:

* under the age of 21 and older than 80
* pregnant
* Type 1 diabetes or diabetes secondary to other conditions
* malignancy or life threatening illness with life expectancy of <5 years
* inability to perform unsupervised physical activity
* diagnosed cognitive deficits or limited decision-making capacity

Provider Surveys Inclusion criteria

* clinicians who are unable to complete the survey in the English language.

Key Informant Interviews Inclusion criteria

* who are unable to participate in the interview conducted in the English language.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Islam, Principal Investigator — NYU Langone
Locations (1):
- NYU Langone, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Researchers who provide a methodologically sound proposal. Upon reasonable request Requests should be directed to laura.wyatt@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Result] Shah MK, Wyatt LC, Gibbs-Tewary C, Zanowiak JM, Mammen S, Islam N. A Culturally Adapted, Telehealth, Community Health Worker Intervention on Blood Pressure Control among South Asian Immigrants with Type II Diabetes: Results from the DREAM Atlanta Intervention. J Gen Intern Med. 2024 Mar;39(4):529-539. doi: 10.1007/s11606-023-08443-6. Epub 2023 Oct 16. PMID 37845588
- [Result] Shah MK, Wyatt LC, Gibbs-Tewary C, Zanowiak J, Mammen S, Mohsin FM, Islam N. Protocol and baseline characteristics for a community health worker-led hypertension and diabetes management program for South Asians in Atlanta: The DREAM Atlanta study. Contemp Clin Trials. 2022 Sep;120:106864. doi: 10.1016/j.cct.2022.106864. Epub 2022 Aug 5. PMID 35940551

RESULTS

PARTICIPANT FLOW:
Groups:
- Non Randomized: Participants who were consented but were not randomized to either group.
Period: Overall Study
Arm/Group | Community Health Workers (CHW) Treatment Group | Control Group | Non Randomized
Started | 97 | 93 | 5
Completed | 92 | 91 | 0
Not Completed | 5 | 2 | 5
Not completed — Lost to Follow-up | 1 | 2 | 0
Not completed — Health Issues | 1 | 0 | 0
Not completed — Left the country | 1 | 0 | 0
Not completed — Unable to maintain time commitment | 1 | 0 | 0
Not completed — No longer interested | 1 | 0 | 0
Not completed — Ineligible post consent | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Population: Baseline data was not collected for the "Non Randomized" Arm/Group as these patients became ineligible post consent, and were removed from the study prior to being randomized to an arm. Only baseline data was reported for the participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Community Health Workers (CHW) Treatment Group | Control Group | Total
Number analyzed (Participants) | 92 | 91 | 183
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (12.5) | 55.8 (11.0) | 56 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 50 | 103
  Male | 39 | 41 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 92 | 91 | 183
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 92 | 91 | 183
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 92 | 91 | 183

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Achieve Blood Pressure (BP) Control.
Description: The primary outcome will be the percentage of eligible patients at a practice site to achieve BP control (130/80 mmHg) six months following the index office visit. The primary outcome will be measured by the treatment participants and providers surveys.
Time Frame: Month 6
Measure: Number; unit: percentage of participants
Arm/Group | Community Health Workers (CHW) Treatment Group | Control Group
Number analyzed (Participants) | 92 | 91
percentage of participants | 40.2 | 24.2

2. Secondary Outcome: Change in Haemoglobin A1c (HbA1c)
Description: Change in HbA1c will be measured in participants of CHW intervention versus the control participants. Clinical data will be retrieved from EHR.
Time Frame: 6 months
Population: This study was launched during COVID and the study team had difficulty collecting the data from all participants due to the pandemic. Data collection from all participants was not an option due to the preference for telemedicine appointments vs in-person appointments. A1c data was collected through the electronic medical record and reported on data that was available, the remaining data is missing.
Measure: Mean (Standard Deviation); unit: Percentage change in HbA1c
Arm/Group | Community Health Workers (CHW) Treatment Group | Control Group
Number analyzed (Participants) | 28 | 19
Percentage change in HbA1c | 6.7 (0.8) | 6.9 (0.9)

3. Secondary Outcome: Systolic Blood Pressure (SBP)
Description: SBP will be measured in participants of CHW intervention versus the control participants. Clinical data will be retrieved from EHR.
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Community Health Workers (CHW) Treatment Group | Control Group
Number analyzed (Participants) | 92 | 91
mmHg | 126.1 (11.3) | 132.5 (12.4)

4. Secondary Outcome: Diastolic Blood Pressure (DBP)
Description: DBP will be measured in participants of CHW intervention versus the control participants. Clinical data will be retrieved from EHR.
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Community Health Workers (CHW) Treatment Group | Control Group
Number analyzed (Participants) | 92 | 91
mmHg | 76.8 (9.2) | 81.0 (7.4)

5. Secondary Outcome: Body Mass Index (BMI)
Description: BMI will be measured in participants of CHW intervention versus the control participants. Clinical data will be retrieved from EHR.
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Community Health Workers (CHW) Treatment Group | Control Group
Number analyzed (Participants) | 92 | 91
kg/m2 | 26.8 (4.5) | 26.7 (4.4)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Community Health Workers (CHW) Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/91
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/91
Other Adverse Events (participants affected / at risk) | 0/92 | 0/91

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/11/NCT04263311/Prot_SAP_000.pdf